CLINICAL TRIAL: NCT02629458
Title: A Study to Determine the Feasibility and Acceptability of Conducting a Phase III Randomised Controlled Trial Comparing Stereotactic Ablative Radiotherapy (SABR) With Surgery in paTients With Peripheral Stage I nOn-small Cell Lung Cancer (NSCLC) cOnsidered Higher Risk of Complications From Surgical Resection
Brief Title: A Study to Determine the Feasibility and Acceptability of Conducting a Phase III Randomised Controlled Trial Comparing Stereotactic Ablative Radiotherapy With Surgery in paTients With Peripheral Stage I nOn-small Cell Lung Cancer cOnsidered Higher Risk of Complications From Surgical Resection
Acronym: SABRTOOTHv1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO14/11248
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients requiring surgery (Experimental)
  Interventions: Procedure: Treatment by Surgical resection; Procedure: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Procedure: Treatment by Surgical resection
Procedure: Stereotactic Ablative Radiotherapy (SABR)

SUMMARY:
Stage I non-small cell lung cancer (NSCLC) is curable and surgery is considered the standard of care for fit, good performance status patients. However, a high proportion of patients with stage 1 NSCLC are elderly and/or have medical co-morbidities and are therefore at higher risk of surgical complications. The optimal treatment for these patients is unknown. SABR may be an equally appropriate treatment but this need to be formally assessed. Funded by the NIHR Research for Patient Benefit, SABRtooth is a UK multi-centre, two-group individually randomised controlled feasibility study of patients with peripheral stage I non-small cell lung cancer considered at higher risk from surgery. In total, 54 patients are planned to be recruited from 4 treatment sites and 2 referral sites. This study aims to determine the feasibility and acceptability of performing a largescale definitive randomised phase III trial comparing surgery with stereotactic ablative radiotherapy (SABR). The qualitative substudy is an exploration of the reasons for nonparticipation in the SABRTooth trial. As the two treatments are very different, patients may have a strong preference for either surgery or SABR, or may feel uncomfortable to have a decision between such distinct options taken out of their hands. Understanding why patients choose not to participate or do not take up their treatment allocation will be crucial in demonstrating that recruiting to a larger scale phase III trial is feasible. We will explore what patients, who have declined particpation in the study or who intiailly consented but subsequently fail to take up their randomimsed treatment arm, understand, perceive and feel about, how the SABRTooth trial was presented to them and their expectations of study burden.

ELIGIBILITY:
Inclusion Criteria:

1. Primary tumour characteristics.
2. Peripherally located tumour as defined in the RTOG 0236 study and UK SABR Consortium guidelines. This states that the tumour must be more than 2cm in axial diameter from a major airway.

   * This includes the trachea, carina, right and left main bronchus and extends to the bifurcation of the right upper, right middle, right lower, left upper and left lower lobe bronchioles
3. No evidence of hilar or mediastinal lymph nodes involvement.

   * Any hilar or mediastinal lymph nodes that are either
   * PET positive or >1cm in axial dimension must be sampled by mediastinoscopy, endobronchial ultrasound or oesophageal endoscopic ultrasound and demonstrate negative cytology and/or pathology
4. Local lung cancer MDT consensus opinion that patient is considered suitable for either surgical resection or SABR treatment AND also to be at higher risk complications from surgical resection
5. Age ≥ 18
6. Female patients must satisfy the investigator that they are not pregnant (negative pregnancy test within 72hrs of surgery of day 1 surgery/SABR), or are not of childbearing potential
7. Able and willing to provide written informed consent

Exclusion Criteria:

1. Previous radiotherapy within the planned treatment volume.
2. History of clinically significant diffuse interstitial lung disease
3. Any history of concurrent or previous invasive malignancy that in the opinion of the investigator could impact on trial outcomes
4. Clinical or radiological evidence of metastatic spread
5. History of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements
6. Previous systemic therapies, including targeted and experimental treatments, for their current lung cancer diagnosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Acheivment of a 'steady state' of recruitment. | Rate of recruitment over months 7 to 21.
  Recruitment rate/month over months 7-21 Recruitment rate/month over months 7-21 In order to demonstrate that recruitment targets for the main trial can be met within an adequate timeframe, the key objective of this feasibility study, a 'steady state' of recruitment must be observed. A formal monitoring of recruitment period will begin 6 months after the start of recruitment (allowing a run-in period for set-up), and an average of 3 patients per month must be recruited (randomised) over a consecutive 15 month period (a minimum of 45 patients) in order to demonstrate a 'steady state' of recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elbanna M, Shiue K, Edwards D, Cerra-Franco A, Agrawal N, Hinton J, Mereniuk T, Huang C, Ryan JL, Smith J, Aaron VD, Burney H, Zang Y, Holmes J, Langer M, Zellars R, Lautenschlaeger T. Impact of Lung Parenchymal-Only Failure on Overall Survival in Early-Stage Lung Cancer Patients Treated With Stereotactic Ablative Radiotherapy. Clin Lung Cancer. 2021 May;22(3):e342-e359. doi: 10.1016/j.cllc.2020.05.024. Epub 2020 Jun 2. PMID 32736936
- [Derived] Franks KN, McParland L, Webster J, Baldwin DR, Sebag-Montefiore D, Evison M, Booton R, Faivre-Finn C, Naidu B, Ferguson J, Peedell C, Callister MEJ, Kennedy M, Hewison J, Bestall J, Gregory WM, Hall P, Collinson F, Olivier C, Naylor R, Bell S, Allen P, Sloss A, Snee M. SABRTooth: a randomised controlled feasibility study of stereotactic ablative radiotherapy (SABR) with surgery in patients with peripheral stage I nonsmall cell lung cancer considered to be at higher risk of complications from surgical resection. Eur Respir J. 2020 Nov 12;56(5):2000118. doi: 10.1183/13993003.00118-2020. Print 2020 Nov. PMID 32616595
- See also: Related Info — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-016-0046-2
- See also: ISRCTN registry — https://doi.org/10.1186/ISRCTN13029788